CLINICAL TRIAL: NCT05452577
Title: Clinical Normative Evaluation of Chronic Insomnia Treated by Traditional Chinese Medicine According to Yin Yang Theory and Its Correlation With Circadian Rhythm
Brief Title: Treatment of Chronic Insomnia According to Yin Yang Theory and Its Correlation With Circadian Rhythm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-SR-015
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Chronic Insomnia; Circadian Rhythm; Traditional Chinese Medicine
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Estazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chinese medicine group (Experimental): Participants received Suanzaoren Decoction and Huanglian Wendan Decoction orally twice daily for 4 weeks.
  Subjects who had previously taken Western medicine hypnotics continued to take them, and those who did not take them did not add Western medicine hypnotics.
  Interventions: Drug: Suanzaoren Decoction and Huanglian Wendan Decoction
- Western medicine group (Active Comparator): Participants received Estazolam 1mg tablet orally once daily for 4 weeks.
  Interventions: Drug: Estazolam 1Mg Tab

INTERVENTIONS:
Drug: Suanzaoren Decoction and Huanglian Wendan Decoction — Twice daily. Chinese herbal medicine includes: includes: 25 grams of Suanzaoren, 10 grams of chuanxiong, 30 grams of fushen, 10 grams of Polygala tenuifolia, 10 grams of Pinellia ternata, 12 grams of tangerine peel, 15 grams of Zhuru, 30 grams of forged keel, 30 grams of forged oyster,10 grams of aurantii fructus, 6 grams of coptis chinensis, 30 grams of Albizzia bark.Add or subtract Chinese herbal medicine according to the different clinical manifestations of each patient.
  Other Names: Wild Jujube Seed Decoction and Huanglian Wendan Decoction
  Arms: Chinese medicine group
Drug: Estazolam 1Mg Tab — 1mg tablet once daily
  Other Names: Estazolam; Estazolam Tablets; Estazolam Pill
  Arms: Western medicine group

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Traditional Chinese medicine (TCM) according to Yin Yang theory for treatment of chronic insomnia .

DETAILED DESCRIPTION:
All subjects giving written informed consent. In this multicenter, controlled, prospective cohort study, the outpatient and inpatient chronic insomnia patients' baseline demographic data were collected, including age, gender, education background, and medication history. Venous blood samples were collected and sent to laboratory test for blood routine, and blood biochemistry at Baseline and Week 4. The Pittsburgh sleep quality index (PSQI) was used to assess the patients' sleep quality at baseline and week 4. Objective sleep quality data is assessed by wearing a Sleep wearable devices. The classic Morningness-Eveningness Questionnaire and wearable devices was used to assess the patients' chronotype at baseline and week 4.Subjects who visit the TCM clinic of this project received Suanzaoren Decoction and Huanglian Wendan Decoction orally twice daily for 4 weeks. Add or subtract Chinese herbal medicine according to the different clinical manifestations of each patient. Subjects from TCM clinic who had previously taken Western medicine hypnotics continued taking them, and for those who had not taken before, Western medicine hypnotics shall not be given/prescribed. Subjects who visit the Western medicine clinic of this project received Estazolam 1mg tablet orally once daily for 4 weeks. The participants will have a follow-up visit every two weeks, and the prescription would be adjusted according to the condition of illness.Cessation rate of Western medicine hypnotics was assessed at Month 6.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients or inpatients.
* It conforms to the chronic insomnia diagnosis standard of Chinese adult insomnia diagnosis and treatment guide (2017 Edition).
* Chronic insomnia patients with Yin yang imbalance and Ying Wei Disharmony Syndrome.
* Informed consent, voluntary participation in the study.

Exclusion Criteria:

* Sleep apnea syndrome leads to insomnia.
* Severe depression, suicidal tendency or having committed suicide.
* Pregnant and lactating women.
* It has serious primary heart, liver, lung, kidney, blood or serious diseases affecting its survival, such as: tumor or AIDS, SCR > 1.5n (n is the upper limit of normal value), ALT > 2n (n is the upper limit of normal value), WBC < 3.0 × 109 / L;
* Those who cannot give full informed consent due to mental disorders.
* According to the researcher's judgment, other situations that are not suitable for the group, such as the change of working environment.
* Subjects who are participating in other clinical studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the total score of the Pittsburgh sleep quality index (PSQI) at 4 weeks | Baseline and Week 4
  The Pittsburgh sleep quality index (PSQI) is a validated,self-reported instrument assessing the sleep quality over the past 4 week period. Possible scores range from 0(the best sleep quality) to 21(the worst possible sleep) quality).The higher the score of PSQI, the worse the sleep quality. Change=(Month 1 Score-Baseline Score)
Cessation rate of Western medicine hypnotics at Month 6 | Month 6
  Cessation was defined as an absence of any Western medicine hypnotics that was sustained for 3 consecutive months or more. Cessation rate of Western medicine hypnotics=(Month 6 number-Baseline number)/Baseline number of Participants use Western medicine hypnotics.

SECONDARY OUTCOMES:
Change from Baseline of the ALT at 4 weeks | Baseline and Week 4
  Alanine aminotransferase, ALT in U/L
Change from Baseline of the AST at 4 weeks | Baseline and Week 4
  Aspartate aminotransferase, AST in U/L
Change from Baseline of the BUN at 4 weeks | Baseline and Week 4
  Blood urea nitrogen, BUN in mmol/L
Change from Baseline of the Scr at 4 weeks | Baseline and Week 4
  Serum creatinine, Scr in μmol/L
Genome-wide association study | Month 6
  Illumina HumanHap550-Duo BeadChips was used to perform the whole genome genotyping in deCODE genetics(Reykjavı'k, Iceland)
Change from Baseline in the score of Morningness-Eveningness Questionaire (MEQ) | Baseline and Week 4
  The MEQ is a validated, self-reported questionaire assessing personal chronotype in the recent period. Possible scores range from 16 (extreme eveningness) to 86 (extreme morningness). Change = (Week 4 Score - Baseline Score). Positive score change indicates a shift from eveningness to morningness.
Change from baseline objective sleep quality | Baseline and Week 4
  Objective sleep quality data is assessed by wearing a Sleep wearable devices

CONTACTS AND LOCATIONS:
Overall Officials: Xiuqin Wang, doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No